CLINICAL TRIAL: NCT05135234
Title: Adaptive Effects of Very Light Physical Activity on Metabolism
Brief Title: Developing a Physiological Understanding of High Duration Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Houston (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Marc Hamilton, Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15463-01; University of Houston (Other Grant/Funding Number: University of Houston)
Record Dates: First submitted 2019-04-16; First posted 2021-11-26 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Sedentary Lifestyle; Hyperinsulinemia; Glucose Tolerance Impaired; Low-density-lipoprotein-type; Aging Problems; Lipid Metabolism Disorders; Inactivity, Physical; Metabolic Disorder, Glucose
Keywords: sedentary; physical activity; muscle contractile activity
MeSH Terms: conditions — Sedentary Behavior; Hyperinsulinism; Glucose Intolerance; Lipid Metabolism Disorders; Glucose Metabolism Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Muscular Exercise (Experimental): Increased level of low effort muscular activity
  Interventions: Behavioral: Muscular Exercise

INTERVENTIONS:
Behavioral: Muscular Exercise — Sedentary time (muscular inactivity when sitting) will be replaced with low effort muscular activity

SUMMARY:
When muscles are not contracting, the local energy demand by muscle and use of specific fuels used to produce energy by oxidative metabolism are minimal. The time people spend sitting inactive (sedentary time) typically comprises more than half of the day. This sedentary behavior is associated with elevated risk of diabetes, cardiovascular diseases, some cancers, and multiple conditions leading to poor aging.

From a progressive series of experiments, the driving goal is to develop a physiological method for sustaining contractile activity via oxidative metabolism over more time than is possible by traditional exercise (hours, not minutes per day).

Developing a physiological method suitable of prolonged muscular activity for ordinary people (who are often unfit) requires gaining fundamental insights about muscle biology and biomechanics. This also entails a careful appreciation of the ability to isolate specific muscles in the leg during controlled movements, such as the soleus muscle during isolated plantarflexion. This includes quantifying specific biological processes that are directly responsive to elevated skeletal muscle recruitment. The investigators will focus on movement that is safe and practical for ordinary people to do given their high amount of daily sitting time.

This includes developing methods to optimally raise muscle contractile activity, in a way that is not limited by fatigue, and is feasible throughout as many minutes of the day as possible safely. This also requires development of methodologies to quantify specific muscular activity, rather than generalized body movement.

There is a need to learn how much people can increase muscle metabolism by physical activity that is perceived to them as being light effort. It is important to learn if this impacts systemic metabolic processes under experimental conditions over a short term time span in order to avoid confounding influences of changes in body weight or other factors.

DETAILED DESCRIPTION:
Physical activity/inactivity will be carefully measured with objective devices. Wearable devices most commonly include accelerometers capable of capturing various types of movement and body posture. The intensity of muscle activation (the soleus and other leg muscles) will be measured in some participants in the developmental studies with EMG, with the limb motion quantified with goniometry. Skeletal muscle and whole body metabolism will be evaluated, especially after isolated local contractile activity focusing on the slow oxidative soleus muscle. Blood chemistry will also be investigated in this comprehensive series of studies to understand how replacing sedentary time with low effort muscular activity can be enhanced. Glycemia will be evaluated in the postprandial period in the morning after an overnight fast when there can be standardized control of carbohydrate ingestion. This includes a standardized oral glucose tolerance test with careful experimental assessment of posture and muscular recruitment during the testing periods. One phase of this study is particularly interested in assessing the acute responses that occur immediately as a result of contractile activity, while also evaluating in another phase how this may be impacted by a change in the sedentary lifestyle. This includes assessing new approaches for improving metabolism throughout the day by reducing the amount of time sitting inactive (i.e. sedentary time). Importantly, because the potential immediate benefits of muscle contractile activity are directly dependent on the duration of activity, the investigators aim to develop in a series of experiments how much muscular activity time can be performed comfortably and safely by anybody instead of sitting inactive with low muscle metabolism regardless of age, fitness, body type, and other conditions commonly limiting effectiveness of traditional exercise prescriptions.

ELIGIBILITY:
Inclusion Criteria:

* Age must be 18 years or older
* Able to fast overnight
* Can maintain diet, medications, and sleep habits between each of the testing visits.
* Lifestyle is consistent with participation in a study evaluating reductions of inactivity (defined by sitting at a low metabolic rate because of minimal muscular activity)
* Willing and able to wear small wearable activity monitors under their clothes as instructed.
* No plans to start a new diet or exercise program if enrolled in the present study.

Exclusion Criteria:

* Practical barriers to completing the study, such as plans to move, or work, or family commitments.
* Plans to change lifestyle during the present study.
* Have physical, vocational, or reasons that prohibit ordinary sitting behaviors present in the modern world.
* Currently dieting to change body weight, or have eating disorder.
* Are pregnant or plan to become pregnant.
* Taking medications that affect bleeding (ie anticoagulants).
* Allergy to lidocaine excludes biopsy component of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Oxygen cost of isolated muscle contractions | Acute contractile activity (at least 3 minutes)
  The energetics of isolated muscle contractions will be described relative to the distinct biomechanics of different types of muscular movement
Fatigue time during muscle group specific contractile activity | Acute measurements less than 1 day. The exact duration is an individual response that is an outcome of unknown minutes consistent with the fatiguability of different movements.
  Determinants of muscular endurance as a function of recruitment intensity
Change in postprandial glucose regulation | The change through the completion of the postprandial period, an average of 180 minutes
  Glucose concentration response during the postprandial period after an oral glucose tolerance test
Change in very low density lipoprotein (VLDL) - Triglyceride | The change through the completion of an acute fasting period, approximately 8-12 hours
  The concentration of triglyceride in the plasma VLDL lipoprotein
The change in muscular inactivity time as a result of isolated contractile activity of the soleus | Throughout the waking day (~16 hours).
  Development of an objective method(s) to quantify sedentary vs. non sedentary time.
Angiopoietin-like protein 4 | The acute time course during the onset of muscular inactivity and contractile activity within 30 minutes to 8 hours
  One of the molecular determinants of lipoprotein lipase regulation

SECONDARY OUTCOMES:
Recruited mass of the soleus and other muscles in the triceps surae during isolated plantarflexion | During acute contractile activity of at least 3 minutes
  grams of the soleus, lateral gastrocnemius and medial gastrocnemius
Electrical activity of muscle, Electromyography (EMG) | At least 3 minute recording periods
  The activation of the triceps surae muscle group
Local rate of oxygen consumption of working muscle | Steady-state measurements taken for ~6 continuous minutes of contractile activity
  oxygen cost per kg muscle during isolated contractile activity and treadmill exercise
The ratio of carbohydrate vs. fat oxidation | Acute responses within less than 24 hours.
  The change in the ratio of the fat vs. carbohydrate utilization during acute contractile activity
Plasma insulin change | The change through the completion of the postprandial period, an average of 180 minutes
  Plasma insulin concentration
Sedentary/muscular inactivity time vs. intermittent non-seated standing behaviors | Throughout the waking day (~16 hours).
  Sedentary time is defined as sitting with a low rate of muscle metabolism due to inactivity
apolipoprotein B100 concentration change | After at least 4 weeks of increased contractile activity
  Biochemical measurement in units of mg per dL
Change in the concentration of GlycA (this is not an acronym; it is a biomarker of inflammation) | After at least 4 weeks of increased contractile activity
  Nuclear magnetic resonance in units of umol per L
Small dense LDL concentration change | After at least 4 weeks of increased contractile activity
  This is an atherogenic lipoprotein particle
Complement component 3 (C3) concentration change | After at least 4 weeks of increased contractile activity
  This is an acute phase protein, a marker of inflammation
Ferritin concentration change | After at least 4 weeks of increased contractile activity
  This is a biomarker related to inflammation and diabetes
Plasma triglyceride concentration change | After at least 4 weeks of increased contractile activity
  Triglyceride concentration in VLDL and non-VLDL particles

CONTACTS AND LOCATIONS:
Overall Officials: Marc T Hamilton, Ph.D., Principal Investigator — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No